CLINICAL TRIAL: NCT06797583
Title: Transcranial Photobiomodulation Treatment in Patients With Sickle Cell Disease
Acronym: PHOTOSCAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PHOTOSCAN
Record Dates: First submitted 2024-12-12; First posted 2025-01-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: The fNIRS device uses light to measure blood flow and oxygen levels in the brain. Participants will be assigned to receive transcranial photobiomodulation or a sham condition using a randomized block design. Randomized block design involving 2 (TPBM): 1(sham) randomization. One group will wear fNIRS headset which will deliver light therapy; or a headset with placebo (no light therapy) and complete a series of computer tests while wearing the headset for 10 minutes. The groups will be divided by genotype (SS/SB0 and SC/SB+) and age (8-12 and 13-17) such that there will be four subgroups that are randomly assigned.
Who Masked: Participant
Masking Description: Research participants will be told of their assigned group (sham control or intervention) after all study procedures are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCD Genotype SS/SB0; Age 8-12 Years (Active Comparator): Transcranial photobiomodulation (TPBM), a light-based treatment using a fNIRS headset to capture changes in cerebral hemodynamics in the prefrontal cortex associated with (TPBM).
  Interventions: Device: Active Transcranial Photobiomodulation (TPBM)
- SCD Genotype - SS/SB0; Age 13-17 Years (Active Comparator): Transcranial photobiomodulation (TPBM), a light-based treatment using a fNIRS headset to capture changes in cerebral hemodynamics in the prefrontal cortex associated with (TPBM).
  Interventions: Device: Active Transcranial Photobiomodulation (TPBM)
- SCD Genotype - SC/SB+; Age 8-12 Years (Sham Comparator): Sham condition using a randomized block design involving 2 (TPBM): 1(sham) randomization.
  Interventions: Device: Sham Transcranial photobiomodulation (TPBM)
- SCD Genotype - SC/SB+; Age 13-17 Years (Sham Comparator): Sham condition using a randomized block design involving 2 (TPBM): 1(sham) randomization.
  Interventions: Device: Sham Transcranial photobiomodulation (TPBM)

INTERVENTIONS:
Device: Active Transcranial Photobiomodulation (TPBM) — CytonBrite, 1064nm LED
  Arms: SCD Genotype - SS/SB0; Age 13-17 Years; SCD Genotype SS/SB0; Age 8-12 Years
Device: Sham Transcranial photobiomodulation (TPBM) — Sham condition using a randomized block design involving 2 (TPBM): 1(sham) randomization.
  Arms: SCD Genotype - SC/SB+; Age 13-17 Years; SCD Genotype - SC/SB+; Age 8-12 Years

SUMMARY:
Participants are being asked to take part in this clinical trial, a type of research study, because investigators want to learn more about oxygen usage in the brain. Patients diagnosed with sickle cell disease are at risk for difficulties with thinking and academic skills. The brain requires a consistent supply of oxygen for normal function, but this supply is reduced among patients with sickle cell disease. The development of new treatments to improve cerebrovascular functioning is needed to limit these difficulties. Transcranial photobiomodulation (i.e., light stimulation to the brain) has the potential to improve cerebrovascular and neurocognitive functioning among patients with sickle cell disease.Participants will be selected randomly (like the flip of a coin) to receive either active light therapy or placebo (no active light treatment).

Primary Objectives

* Measure the participation rate in a study of transcranial photobiomodulation to improve cognitive functioning in a sample of children with sickle cell disease (ages 8- 17 years).
* Assess self- and caregiver-reported ratings of feasibility and acceptability.
* Evaluate the frequency and nature of side effects associated with transcranial photobiomodulation.

Secondary Objectives

* To assess the change in cognitive performance associated with transcranial photobiomodulation compared to a sham control condition.
* To measure changes in cerebrovascular oxygenation (oxygenated and deoxygenated hemoglobin) following transcranial photobiomodulation compared to a sham control condition.

DETAILED DESCRIPTION:
Patients diagnosed with sickle cell disease (SCD) of any genotype, between the ages of 8-17 years will be recruited through the Sickle Cell Clinical Research and Intervention Program (SCCRIP). Recruited participants will be selected randomly to receive TPBM (CytonBrite, 1064nm LED) or a sham condition using a randomized block design involving 2 (TPBM): 1(sham) randomization. The groups will be divided by genotype (SS/SB0 and SC/SB+) and age (8-12 and 13-17) such that there will be four subgroups that are randomly assigned.

Participants will be asked to complete a baseline side effects questionnaire (modified Patient Report of Incidence of Side Effects and Visual Analog Pain Scale) and caregivers will complete a medical/demographics questionnaire.

After completing the baseline questionnaires, a functional near infrared spectroscopy (fNIRS) headband (NIRSport2) will be fitted for the participant based on the circumference of their head. The cap is then fitted with emitters and detectors to capture changes in cerebral hemodynamics in the frontal cortex.

Prior to wearing the headband, participants will complete an assessment to estimate overall intellectual abilities based on their vocabulary skills (NIH Picture Vocabulary Test). Then the participants will complete four cognitive measures associated with frontal functioning while wearing the fNIRS headband. These tasks measure processing speed and working memory and take approximately 5-6 minutes each to complete.

Photobiomodulation using the CytonBrite PBM device will be performed immediately following the initial fNIRS exam. The CytonBrite headpiece will be placed on the head. The six LED probes will be positioned over the forehead, and the probes will be adjusted per device specifications to maximize light penetration to the prefrontal cortex. The patient will receive 10 minutes of continuous wave light or sham.

Following stimulation or sham, the fNIRS cap will be placed in the same location and the same cognitive measures will be completed (4 measures of frontal functioning). Changes in cerebral hemodynamics and cognitive performance on four measures (2 working memory and 2 processing speed tasks) from pre- to post-stimulation will be compared between the two groups. This will take about 30 minutes.

The cap will be removed, and the caregiver and the participant will complete brief rating forms assessing perceived feasibility and acceptability of the intervention (FIM and AIM). Additionally, participants will be asked to report any side effects they experienced immediately following the intervention.

Among the participants that were randomized to TPBM, the sample (both caregiver and participant) will be further randomized to complete a brief (~10-15 minutes) interview assessing the perceived feasibility and acceptability of the TPBM intervention.

Approximately one-week post-intervention, participants will complete the side effects questionnaires virtually.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with sickle cell disease of any genotype
* Enrolled in the Sickle Cell Clinical Research and Intervention Program (SCCRIP)
* Between the ages of 8 to 17 years
* Primary language is English
* Participant and Parent/Legal Guardian is willing to participate and provide consent/assent according to institutional guidelines

Exclusion Criteria:

* History of an abnormal transcranial doppler screening
* History of a documented silent cerebral infarct
* History of documented central nervous system injury, including a traumatic brain injury, Moya Moya disease, or overt stroke
* Participant received transfusion treatment within the past three months.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Measure the participation rate in a study of transcranial photobiomodulation to improve cognitive functioning in a sample of children with sickle cell disease (ages 8-17 years). | Through study completion of all enrolled participants, estimated to be 3 years
  A binary variable indicating whether a participant engaged in the study (1 = participated, 0 = did not participate). Overall participation rate will be calculated as the proportion of participants who engaged in this study.
Assess self-reported ratings of feasibility. | Immediately post intervention period
  Subgroup analysis and logistic regression analysis will be used to describe factors of interest which may impact participation rates.
Assess self-reported ratings of acceptability. | Immediately post intervention period
  Subgroup analysis and logistic regression analysis will be used to describe factors of interest which may impact participation rates.
Assess caregiver-reported ratings of feasibility. | Immediately post intervention period
  Subgroup analysis and logistic regression analysis will be used to describe factors of interest which may impact participation rates. Qualitative metrics will also be used to analyze semi-structured interviews.
Assess caregiver-reported ratings of acceptability. | Immediately post intervention period
  Subgroup analysis and logistic regression analysis will be used to describe factors of interest which may impact participation rates. Qualitative metrics will also be used to analyze semi-structured interviews.
Evaluate the frequency and nature of side effects associated with transcranial photobiomodulation. | Immediately before intervention, immediately after intervention and one week post intervention period.
  The frequency and percentage of each type of side effect will be calculated along with summary statistics for the nature and frequency of side effects.
Evaluate the frequency and nature of side effects associated with transcranial photobiomodulation. | Immediately before intervention, immediately after intervention and one week post intervention period
  Descriptive statistics of self-report ratings on the Visual Analog Pain Scale will be reported.

SECONDARY OUTCOMES:
To assess the change in cognitive performance associated with transcranial photobiomodulation | Assessed immediately before and immediately after intervention.
  For each subject's cognitive performance in both sessions of the psychomotor vigilance task (PVT) and delayed match to sample (DMS) task, an overall cognitive score will be calculated, incorporating both speed (reaction time) and accuracy (number of correct responses), using the rate correct score. This overall cognitive score is equal to the number of correct responses divided by the sum of all reaction times. The behavioral results for all 4 cognitive measures will be analyzed with an independent two-sample t-test comparing performance on these tasks before and after stimulation for two groups with a one-tailed level of significance with p ≤ 0.10.
To assess the change in cognitive performance associated with transcranial photobiomodulation. | Assessed immediately before and immediately after intervention
  Age-standardized scores for the NIH Toolbox List Sorting and NIH Toolbox Pattern Comparison test will be calculated. The behavioral results for all 4 cognitive measures will be analyzed with an independent two-sample t-test comparing performance on these tasks before and after stimulation for two groups with a one-tailed level of significance with p ≤ 0.10.
To assess the change in cognitive performance associated with a sham control condition. | Assessed immediately before and immediately after intervention.
  For each subject's cognitive performance in both sessions of the psychomotor vigilance task (PVT) and delayed match to sample (DMS) task, an overall cognitive score will be calculated, incorporating both speed (reaction time) and accuracy (number of correct responses), using the rate correct score. This overall cognitive score is equal to the number of correct responses divided by the sum of all reaction times. The behavioral results for all 4 cognitive measures will be analyzed with an independent two-sample t-test comparing performance on these tasks before and after stimulation for two groups with a one-tailed level of significance with p ≤ 0.10.
To assess the change in cognitive performance associated with a sham control condition. | Assessed immediately before and immediately after intervention
  Age-standardized scores for the NIH Toolbox List Sorting and NIH Toolbox Pattern Comparison test will be calculated. The behavioral results for all 4 cognitive measures will be analyzed with an independent two-sample t-test comparing performance on these tasks before and after stimulation for two groups with a one-tailed level of significance with p ≤ 0.10.
To measure changes in cerebrovascular oxygenation (oxygenated and deoxygenated hemoglobin) following transcranial photobiomodulation. | Assessed immediately before and immediately after intervention.
  Means will be calculated for HbO2 and Hb levels in each group. Hypothesis tests will be conducted to determine if there are statistically significant differences in HbO2 and Hb levels between the treatment and control groups. Appropriate parametric or non-parametric tests will be utilized based on data distribution and assumptions. The effect sizes (e.g., Cohen's d) will also be calculated to quantify the magnitude of the differences observed.
To measure changes in cerebrovascular oxygenation (oxygenated and deoxygenated hemoglobin) following a sham control condition. | Assessed immediately before and immediately after intervention.
  Meanswill be calculated for HbO2 and Hb levels in each group. Hypothesis tests will be conducted to determine if there are statistically significant differences in HbO2 and Hb levels between the treatment and control groups. Appropriate parametric or non-parametric tests will be utilized based on data distribution and assumptions. The effect sizes (e.g., Cohen's d) will also be calculated to quantify the magnitude of the differences observed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Heitzer, PhD, Principal Investigator — St. Jude Children's Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the ClinicalTrials.gov (CTG) website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols